CLINICAL TRIAL: NCT02824666
Title: Phase 1, Open-Label Positron Emission Tomography (PET) Study to Evaluate D2 Receptor Occupancy Following Single Intravenous Administration of ATI-9242 in Adult Male Healthy Subjects
Brief Title: Study to Evaluate D2 Receptor Occupancy Following Single Intravenous Administration of ATI-9242
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Braeburn Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BB-ATI9242-001
Record Dates: First submitted 2016-06-08; First posted 2016-07-07 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5 mg/kg (Experimental): • Cohort 1: ATI-9242 - Single IV bolus dose of 0.5 mg/kg
  Interventions: Drug: ATI-9242; Radiation: [18F]Fallypride Imaging
- ATI-9242 1.0 mg/kg (Experimental): • Cohort 2: ATI-9242 - Single IV bolus dose of 1.0 mg/kg
  Interventions: Drug: ATI-9242; Radiation: [18F]Fallypride Imaging

INTERVENTIONS:
Drug: ATI-9242 — Formulated ATI-9242 will be administered as an IV bolus injection (2mg/mL of ATI-9242 in 40% solution of propylene glycol).
  Two doses will be tested: single IV bolus injection of 0.5mg/kg and single IV bolus injection 1.0 mg/kg. In the event that a third cohort is needed the IV bolus injection would be 2.0 mg/kg
Radiation: [18F]Fallypride Imaging — Subjects will be injected with approximately 250 MBq or 6.75 mCi of [18F]Fallypride [5-6 mCi being the typical range of injected dose].

SUMMARY:
This study involves evaluating the occupancy of ATI-9242 at steady state at three different dose levels on D2 receptors in the brain using [18F] Fallypride PET in up to three cohorts of subjects.

DETAILED DESCRIPTION:
This study involves evaluating the occupancy of ATI-9242 at steady state at three different dose levels on D2 receptors in the brain using [18F]Fallypride PET in up to three cohorts of subjects. The first dose evaluated will be 0.5 mg/kg administered as an IV bolus injection. The second dose that will be evaluated will be 1.0 mg/kg as an IV bolus injection. The safety and occupancy after each dose level will be evaluated prior to moving to the next dose. On two separate days, subjects will undergo [18F]Fallypride PET imaging sessions. The plasma concentration of ATI-9242 will be obtained prior to and during the course of the imaging session to allow determination of the relationship between plasma concentration of ATI-9242 with in vivo D2 occupancy.

ELIGIBILITY:
Inclusion Criteria:

* Are males > 18 years of age and < 50 years of age.
* BMI <30
* Are in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
* Are able to communicate well with the investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent.
* Provide informed consent for study procedures.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects and for 90 days after the end of the study.
* Subjects must not donate sperm for the study duration and for 90 days after the end of the study.
* Willing and able to cooperate with study procedures
* A brain MRI within the past 120 days with no evidence of active or focal neurological disease that may interfere with the [18F]Fallypride PET data.

Exclusion Criteria:

* Use of any prescription drugs, herbal supplements, within four (4) weeks prior to Baseline imaging, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to Baseline imaging. If needed (i.e. an incidental and limited need), acetaminophen is acceptable, but must be documented as a concomitant medication/significant non-drug therapy.
* Exposure to any investigational drug within the 4 weeks prior to screening visit.
* Subjects with a history of exposure to any radiation >15 mSv/year (e.g., occupational or radiation therapy) over the past year.
* Donation or loss of 400 ml or more of blood within eight (8) weeks prior to initial dosing, or longer if required by local regulation.
* Have a history or presence of any significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders which, in the opinion of the investigator, are capable of altering the absorption, metabolism, or elimination of drugs or posing a health risk to participate in the study.
* Have clinically significant findings on laboratory evaluations in the opinion of the investigator.
* Have clinically significant findings on ECG evaluation.
* A positive Hepatitis B surface antigen (HBsAg), Hepatitis C antibody or HIV test result.
* History of drug or alcohol abuse within the 12 months prior to screening, or evidence of such abuse as indicated by the laboratory assays conducted during the screening.
* History of tobacco product use within 3 months prior to screening, to be verified by urine cotinine screening.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI.
* Claustrophobia that would interfere with completion of MRI and/or SPECT procedures.
* Inability to lie supine for 90 minutes at a time.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-09-06 (Actual); Study Completion 2016-11-08 (Actual)

PRIMARY OUTCOMES:
Target receptor occupancy after single intravenous(IV) of ATI-9242 in 6 healthy adults using the D2 receptor ligand [18F]Fallypride and PET imaging. | approximately 5 weeks
  Change from baseline in PET imaging at baseline of ATI-9242 and post-dose

SECONDARY OUTCOMES:
Explore the relationship between ATI-9242 dose, plasma concentrations of ATI-9242 and target receptor occupancy in 6 subjects. | approximately 5 weeks
  The relationship between plasma drug concentration/PK parameters of ATI-9242 and D2 occupancy will be explored.

OTHER OUTCOMES:
Safety and tolerability of ATI-9242 following single IV dose in 6 healthy subjects via safety assessments . | approximately 5 weeks
  incidence of adverse events (AEs), vital signs (blood pressure, pulse and oral temperature), physical examinations 12-lead ECG, CSSRS and clinical laboratory tests (hematology, clinical chemistry and urinalysis).

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana Clinical Research Center, IU Health University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No